CLINICAL TRIAL: NCT04436679
Title: INTER-Regional COHORTE of Long Term Pancreatic Cancer Survivors
Acronym: CaPaLong
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_29; 2019-A02001-56 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pancreas Cancer; Pancreatic Adenocarcinoma
Keywords: survival; prognosis; tissue; pancreas cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissues paraffin lumbered paraffin blocks of tissue-microarrays
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is particularly innovative as it will accurately analyze the microscopic characteristics of the stroma, tumor budding and mucin expression in adenocarcinomas of the pancreas, using a comparative approach of long-survivor/short-survival patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age at diagnosis
* Primary pancreatic cancer patients operated on in one of the 4 centres between 2001 and 2016
* Histopathological diagnosis of excreto-pancreatic adenocarcinoma of the pancreas, ductal adenocarcinoma or classical adenocarcinoma
* Tissue blocks (FFPE) available (tumour/healthy tissue)
* Affiliated to a social security scheme

Exclusion Criteria:

* Absence of Primary Cancer Tissue Blocks (PCTBs)
* Paraffin block fixed in Bouin or AFA
* Patient Refusal
* Pancreatic cancer not corresponding to a conventional excretopancreatic adenocarcinoma such as: carcinoma on intraductal papillary mucinous neoplasm, endocrine tumor/carcinoma, acinar cell carcinoma, ...).
* Patient died due to post-surgical complications (death within 30 days post-surgery).
* Surgical resection of macroscopic R2 type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic adenocarcinoma patients operated on between 2001 and 2016.
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Relationship between known prognostic histological markers of pancreatic adenocarcinoma and patient survival. | at 2 years
  Tissue analysis will be performed by conventional microscopy and will evaluate histological markers known in the literature to have a prognostic impact.

SECONDARY OUTCOMES:
Relationship between newly described histological markers for pancreatic adenocarcinoma and patient survival. | at 2 years
  Immunohistochemistry tissue analysis. It will allow the evaluation of newly described histological markers for pancreatic adenocarcinoma, which could have a prognostic impact such as the immunophenotype of the inflammatory infiltrate, the expression of the mucins MUC1, MUC5AC, MUC4, MUC16, mesothelin, p53, Ki67 (MIB1) and markers of aggressive subtypes identified by transcriptome studies, in particular the basal-like molecular subtype.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Leteurtre, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France